CLINICAL TRIAL: NCT04715581
Title: Effect of Multicomponent Prehabilitation on Early and Long-term Outcomes in Elderly Patients With Frailty After Digestive Surgery for Cancer: A Randomized-controlled Study
Brief Title: Multicomponent Prehabilitation and Outcomes in Elderly Patients With Frailty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2020-331
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Old Age; Debility; Digestive Cancer; Surgery; Preoperative Rehabilitation; Nutrition Therapy; Outcomes
Keywords: older patients; frailty; digestive cancer; prehabilitation; nutrition therapy; outcomes
MeSH Terms: conditions — Frailty; Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent prehabilitation group (Experimental): Patients in the intervention group will receive nutritional optimization and exercise training before the surgery, exercise training after the surgery, and home-based rehabilitation after discharge.
  Interventions: Dietary Supplement: Preoperative nutritional optimization; Behavioral: Preoperative exercise training; Behavioral: Postoperative exercise training
- Control group (No Intervention): Patients in the control group will maintain normal diet and normal activity before surgery, normal activity after surgery, and normal activity after discharge.

INTERVENTIONS:
Dietary Supplement: Preoperative nutritional optimization — 1. Indication for oral nutritional supplementation: Patients at risk of malnutrition (MNA-SF 8-11) or with malnutrition (MNA-SF 0-7).
  2. Protocol of nutritional optimization: Enteral nutritional powder (Ensure for patients without diabetes and Glucerna for patients with diabetes) twice a day. The target protein intake is 1.5-1.8 g/kg/d. Patients with iron deficient anemia (hemoglobin <130 g/L for men and <120 g/L for women) will be given oral iron therapy.
  3. The duration of nutritional optimization: The day admitted to the hospital to the surgery to one day prior to the surgery.
  Arms: Multicomponent prehabilitation group
Behavioral: Preoperative exercise training — 1. The respiratory training will be performed for at least 2-3 times per day. Respiratory training include thoracic breathing exercise and cough training.
  2. Aerobic exercise will be performed for at least 1-2 times per day. Aerobic exercise includes jogging, walking or climbing stairs. Exercise intensity will be based on patients' tolerance. The goal of the training is to complete the training plan as far as possible.
  3. Every training should be last for 45 minutes to 1 hour. If the patient can not tolerate, the training time should be reduce to 30 minutes.
  4. The duration of exercise training: The day admitted to the hospital to the surgery to one day prior to the surgery.
  Arms: Multicomponent prehabilitation group
Behavioral: Postoperative exercise training — 1. Muscle strength training in the bedside and walking in the ward.
  2. Aerobic exercise includes jogging, walking or climbing stairs. Exercise intensity will be based on patients' tolerance. The goal of the training is to complete the training plan as far as possible.
  3. Exercise training is performed under the supervision of physiotherpists durign hospital stay, and is reminded by regular telephone calls and phone messages after hospital discharge.
  Arms: Multicomponent prehabilitation group

SUMMARY:
The study is designed to investigate the effect of a multicomponent prehabilitation pathway on early and long-term outcomes in elderly patients with frailty recovering from surgery for digestive cancer.

DETAILED DESCRIPTION:
Frailty is an age-related syndrome characterized with diminished physiological reserve that results in decreased homeostatic capacity and increased vulnerability to any stress from minor to major. Approximately 10% to 20% of adults aged 65 years and older present with frailty, and the incidence doubles among those of 85 years and older. Among elderly cancer patients especially those with digestive cancer, the prevalence of frailty and pre-frailty can be as high as 50%. Malnutrition often coexists with frailty, and indeed contribute to the development of frailty. As a matter of fact, the proportion of malnutrition also increases with age even in high-income countries.

Frailty is strongly associated with worsening outcomes in surgical patients, including higher delirium, high non-delirium complications, high perioperative mortality, as well as decreased activity of daily life, cognitive dysfunction and work disability in long-term survivors. Furthermore, malnutrition as a prominent factor in the development of frailty also has adverse impacts on the duration of hospitalization, complications, and survival after surgery. Therefore, it is urgently needed to understand how to enhance the recovery of these patients following surgery.

Exercises and rehabilitation, in combination with nutritional supplement, may reverse or mitigate frailty, promote postoperative recovery, and improve clinical outcomes. However, the reported effectiveness varies with interventions and are not sufficiently robust to guide good clinical practice. The purpose of this study is to investigate the effect of multimodal prehabilitation on early and long-term outcomes in elderly patients with frailty.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥65 years but <90 years;
2. Scheduled to undergo major surgery for digestive cancer with an expected duration of 2 hours and longer, including cancers of esophagus, stomach, small intestine, colon, rectum, pancreas, liver, and biliary tract;
3. Clinical Frailty Scale ≥5;
4. Provide written informed consent.

Exclusion Criteria:

1. Preoperative history of schizophrenia, epilepsy, Parkinsonism, or myasthenia gravis;
2. Inability to communicate due to coma, profound dementia, or language barrier;
3. Inability to participate in preoperative rehabilitation due to paralysis, fracture or other movement disorder;
4. Inability to take oral diet due to preoperative gastrointestinal disease or other disease;
5. Severe heart dysfunction (left ventricular ejection fraction <30% or New York Heart Association classification IV), severe hepatic dysfunction (Child-Pugh class C), severe renal dysfunction (undergoing dialysis before surgery), or American Society of Anesthesiologists classification of grade 4 or higher;
6. Other reasons that are considered unsuitable for study participation.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
A composite of delirium and non-delirium complications within 7 days after surgery (sub-study). | Up to 7 days after surgery.
  Delirium will be assessed with the 3-Dimensional Confusion Assessment Method. Non-delirium complications are defined as new onset medical events other than delirium that are harmful to patients' recovery and required therapeutic intervention, i.e., grade II or higher on Clavien-Dindo classification.
Recurrence-free survival after surgery. | Up to two years after surgery.
  Events include recurrence, metastasis, or all-cause death, whichever come first.

SECONDARY OUTCOMES:
Intensive care unit admission after surgery (sub-study). | Up to 30 days after surgery.
  Intensive care unit admission after surgery.
Incidence of delirium within 7 days after surgery (sub-study). | Up to 7 days after surgery.
  Delirium will be assessed with the 3-Dimensional Confusion Assessment Method.
Time to oral fluid intake after surgery (sub-study). | Up to 30 days after surgery.
  Time to oral fluid intake after surgery.
Time to oral food intake after surgery (sub-study). | Up to 30 days after surgery.
  Time to oral food intake after surgery.
Time to out-of-bed activity after surgery (sub-study). | Up to 30 days after surgery.
  Time to out-of-bed activity after surgery.
6-minute walk distance at hospital discharge (sub-study). | At hospital discharge, up to 30 days after surgery.
  6-minute walk distance at hospital discharge.
Length of hospital stay after surgery (sub-study). | Up to 30 days after surgery.
  Length of hospital stay after surgery.
Incidence of non-delirium complication within 30 days after surgery (sub-study). | Up to 30 days after surgery.
  Non-delirium complications are defined as new onset medical events other than delirium that are harmful to patients' recovery and required therapeutic intervention, i.e., grade II or higher on Clavien-Dindo classification.
All-cause 30-day mortality after surgery (sub-study). | Up to 30 days after surgery.
  All-cause 30-day mortality after surgery.
Quality of life at 30 days after surgery (sub-study). | At 30 days after surgery.
  Quality of life will be assessed with the World Health Organization Quality of Life brief version (WHOQOL-BREF) which is a 24-item questionnaire that assesses the quality of life in physical, psychological, and social relationship, and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.
Cognitive function at 30 days after surgery (sub-study). | At 30 days after surgery.
  Cognitive function will be assessed with the Modified Telephone Interview for Cognitive Status (TICS-m) which is a 12-item questionnaire that verbally assesses global cognitive function via telephone. The score ranges from 0 to 50, with higher score indicating better function.
Sleep quality at 30 days after surgery (sub-study). | At 30 days after surgery.
  Sleep quality will be assessed with the Pittsburgh sleep quality index which is a 9-item questionnaire that assess subjective quality of sleep during the past 1 month. The score ranges from 0 to 21, with higher score indicating poor sleep quality.
Overall survival after surgery. | Up to 2 years after surgery.
  Events include all-cause death.
Cancer specific survival after surgery. | Up to 2 years after surgery.
  Events are cancer-specific death which is defined as death fully attributable to the cancer for which the index surgery is performed and usually involving cancer recurrence and/or metastasis after exclusion of other causes such as stroke and myocardial infarction. Deaths from other causes are censored at the time of death.
Event-free survival after surgery. | Up to 2 years after surgery.
  Events include recurrence/metastasis, new-onset diseases, new-onset tumors, or all-cause mortality, whichever come first.
Physical activity at 30 days after surgery (sub-study). | At 30 days after surgery.
  Physical activity will be assessed with International Physical Activity Questionnaire-Long.

OTHER OUTCOMES:
Intensity of pain after surgery (sub-study). | Up to 7 days after surgery.
  Intensity of pain will be assessed twice daily with the numeric rating scale which is a 11-point scale where 0=no pain and 10=the worst pain.
Subjective sleep quality after surgery (sub-study). | Up to 7 days after surgery.
  Subjective sleep quality will be assessed daily with the numeric rating scale which is a 11-point scale where 0=the best sleep and 10=the worst sleep.
Sleep architecture during the night of surgery (sub-study, part of enrolled patients). | During the night of surgery.
  Sleep will be evaluated with the polysomnographic monitoring during the night of surgery.
Quality of life at 1 year after surgery. | At 1 year after surgery.
  Quality of life will be assessed with the World Health Organization Quality of Life brief version (WHOQOL-BREF) which is a 24-item questionnaire that assesses the quality of life in physical, psychological, and social relationship, and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.
Cognitive function at 1 year after surgery. | At 1 year after surgery.
  Cognitive function will be assessed with the Modified Telephone Interview for Cognitive Status (TICS-m) which is a 12-item questionnaire that verbally assesses global cognitive function via telephone. The score ranges from 0 to 50, with higher score indicating better function.
Serum level of irisin before anesthesia | Intraoperative (Before anesthesia on the day of surgery)
  Blood samples will be collected before anesthesia. Serum will be separated and immediately frozen at -80 °C. Irisin concentration will be measured using a commercial ELISA kit, according to the manufacturer's instructions.
Serum level of irisin on postoperative day 1 | At the first day after surgery
  Blood samples will be collected before anesthesia. Serum will be separated and immediately frozen at -80 °C. Irisin concentration will be measured using a commercial ELISA kit, according to the manufacturer's instructions.
Physical activity at 3 months, 6 months and 1 year after surgery. | At 3 months, 6 months and 1 year after surgery
  Physical activity will be assessed with International Physical Activity Questionnaire-Long.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Collard RM, Boter H, Schoevers RA, Oude Voshaar RC. Prevalence of frailty in community-dwelling older persons: a systematic review. J Am Geriatr Soc. 2012 Aug;60(8):1487-92. doi: 10.1111/j.1532-5415.2012.04054.x. Epub 2012 Aug 6. PMID 22881367
- [Background] Song X, Mitnitski A, Rockwood K. Prevalence and 10-year outcomes of frailty in older adults in relation to deficit accumulation. J Am Geriatr Soc. 2010 Apr;58(4):681-7. doi: 10.1111/j.1532-5415.2010.02764.x. Epub 2010 Mar 22. PMID 20345864
- [Background] Mohile SG, Xian Y, Dale W, Fisher SG, Rodin M, Morrow GR, Neugut A, Hall W. Association of a cancer diagnosis with vulnerability and frailty in older Medicare beneficiaries. J Natl Cancer Inst. 2009 Sep 2;101(17):1206-15. doi: 10.1093/jnci/djp239. Epub 2009 Jul 28. PMID 19638506
- [Background] Verlaan S, Ligthart-Melis GC, Wijers SLJ, Cederholm T, Maier AB, de van der Schueren MAE. High Prevalence of Physical Frailty Among Community-Dwelling Malnourished Older Adults-A Systematic Review and Meta-Analysis. J Am Med Dir Assoc. 2017 May 1;18(5):374-382. doi: 10.1016/j.jamda.2016.12.074. Epub 2017 Feb 24. PMID 28238676
- [Background] Guyonnet S, Rolland Y. Screening for Malnutrition in Older People. Clin Geriatr Med. 2015 Aug;31(3):429-37. doi: 10.1016/j.cger.2015.04.009. Epub 2015 May 13. PMID 26195101
- [Background] Zhang DF, Su X, Meng ZT, Cui F, Li HL, Wang DX, Li XY. Preoperative severe hypoalbuminemia is associated with an increased risk of postoperative delirium in elderly patients: Results of a secondary analysis. J Crit Care. 2018 Apr;44:45-50. doi: 10.1016/j.jcrc.2017.09.182. Epub 2017 Sep 29. PMID 29055835
- [Background] Zhang Y, Shan GJ, Zhang YX, Cao SJ, Zhu SN, Li HJ, Ma D, Wang DX; First Study of Perioperative Organ Protection (SPOP1) Investigators. Preoperative vitamin D deficiency increases the risk of postoperative cognitive dysfunction: a predefined exploratory sub-analysis. Acta Anaesthesiol Scand. 2018 Aug;62(7):924-935. doi: 10.1111/aas.13116. Epub 2018 Mar 26. PMID 29578249
- [Background] Cruz-Jentoft AJ, Kiesswetter E, Drey M, Sieber CC. Nutrition, frailty, and sarcopenia. Aging Clin Exp Res. 2017 Feb;29(1):43-48. doi: 10.1007/s40520-016-0709-0. Epub 2017 Feb 2. PMID 28155181
- [Background] Wei K, Nyunt MSZ, Gao Q, Wee SL, Ng TP. Frailty and Malnutrition: Related and Distinct Syndrome Prevalence and Association among Community-Dwelling Older Adults: Singapore Longitudinal Ageing Studies. J Am Med Dir Assoc. 2017 Dec 1;18(12):1019-1028. doi: 10.1016/j.jamda.2017.06.017. Epub 2017 Aug 10. PMID 28804010
- [Background] Laur CV, McNicholl T, Valaitis R, Keller HH. Malnutrition or frailty? Overlap and evidence gaps in the diagnosis and treatment of frailty and malnutrition. Appl Physiol Nutr Metab. 2017 May;42(5):449-458. doi: 10.1139/apnm-2016-0652. Epub 2017 Mar 21. PMID 28322060
- [Background] Ethun CG, Bilen MA, Jani AB, Maithel SK, Ogan K, Master VA. Frailty and cancer: Implications for oncology surgery, medical oncology, and radiation oncology. CA Cancer J Clin. 2017 Sep;67(5):362-377. doi: 10.3322/caac.21406. Epub 2017 Jul 21. PMID 28731537
- [Background] Lin HS, Watts JN, Peel NM, Hubbard RE. Frailty and post-operative outcomes in older surgical patients: a systematic review. BMC Geriatr. 2016 Aug 31;16(1):157. doi: 10.1186/s12877-016-0329-8. PMID 27580947
- [Background] Fagard K, Leonard S, Deschodt M, Devriendt E, Wolthuis A, Prenen H, Flamaing J, Milisen K, Wildiers H, Kenis C. The impact of frailty on postoperative outcomes in individuals aged 65 and over undergoing elective surgery for colorectal cancer: A systematic review. J Geriatr Oncol. 2016 Nov;7(6):479-491. doi: 10.1016/j.jgo.2016.06.001. Epub 2016 Jun 21. PMID 27338516
- [Background] Richards SJG, Frizelle FA, Geddes JA, Eglinton TW, Hampton MB. Frailty in surgical patients. Int J Colorectal Dis. 2018 Dec;33(12):1657-1666. doi: 10.1007/s00384-018-3163-y. Epub 2018 Sep 14. PMID 30218144
- [Background] Inouye SK, Westendorp RG, Saczynski JS, Kimchi EY, Cleinman AA. Delirium in elderly people--authors'reply. Lancet. 2014 Jun 14;383(9934):2045. doi: 10.1016/S0140-6736(14)60994-6. No abstract available. PMID 24931690
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Persico I, Cesari M, Morandi A, Haas J, Mazzola P, Zambon A, Annoni G, Bellelli G. Frailty and Delirium in Older Adults: A Systematic Review and Meta-Analysis of the Literature. J Am Geriatr Soc. 2018 Oct;66(10):2022-2030. doi: 10.1111/jgs.15503. Epub 2018 Sep 21. PMID 30238970
- [Background] Bellelli G, Moresco R, Panina-Bordignon P, Arosio B, Gelfi C, Morandi A, Cesari M. Is Delirium the Cognitive Harbinger of Frailty in Older Adults? A Review about the Existing Evidence. Front Med (Lausanne). 2017 Nov 8;4:188. doi: 10.3389/fmed.2017.00188. eCollection 2017. PMID 29167791
- [Background] Nomura Y, Nakano M, Bush B, Tian J, Yamaguchi A, Walston J, Hasan R, Zehr K, Mandal K, LaFlam A, Neufeld KJ, Kamath V, Hogue CW, Brown CH 4th. Observational Study Examining the Association of Baseline Frailty and Postcardiac Surgery Delirium and Cognitive Change. Anesth Analg. 2019 Aug;129(2):507-514. doi: 10.1213/ANE.0000000000003967. PMID 30540612
- [Background] Brown CH 4th, Max L, LaFlam A, Kirk L, Gross A, Arora R, Neufeld K, Hogue CW, Walston J, Pustavoitau A. The Association Between Preoperative Frailty and Postoperative Delirium After Cardiac Surgery. Anesth Analg. 2016 Aug;123(2):430-5. doi: 10.1213/ANE.0000000000001271. PMID 27096563
- [Background] Mazzola P, Ward L, Zazzetta S, Broggini V, Anzuini A, Valcarcel B, Brathwaite JS, Pasinetti GM, Bellelli G, Annoni G. Association Between Preoperative Malnutrition and Postoperative Delirium After Hip Fracture Surgery in Older Adults. J Am Geriatr Soc. 2017 Jun;65(6):1222-1228. doi: 10.1111/jgs.14764. Epub 2017 Mar 6. PMID 28263371
- [Background] Ringaitiene D, Gineityte D, Vicka V, Zvirblis T, Sipylaite J, Irnius A, Ivaskevicius J, Kacergius T. Impact of malnutrition on postoperative delirium development after on pump coronary artery bypass grafting. J Cardiothorac Surg. 2015 May 20;10:74. doi: 10.1186/s13019-015-0278-x. PMID 25990791
- [Background] Liu X, Wu X, Zhou C, Hu T, Ke J, Chen Y, He X, Zheng X, He X, Hu J, Zhi M, Gao X, Hu P, Wu X, Lan P. Preoperative hypoalbuminemia is associated with an increased risk for intra-abdominal septic complications after primary anastomosis for Crohn's disease. Gastroenterol Rep (Oxf). 2017 Nov;5(4):298-304. doi: 10.1093/gastro/gox002. Epub 2017 Feb 20. PMID 29230300
- [Background] Ensrud KE, Blackwell TL, Ancoli-Israel S, Redline S, Cawthon PM, Paudel ML, Dam TT, Stone KL. Sleep disturbances and risk of frailty and mortality in older men. Sleep Med. 2012 Dec;13(10):1217-25. doi: 10.1016/j.sleep.2012.04.010. Epub 2012 Jun 15. PMID 22705247
- [Background] Su X, Wang DX. Improve postoperative sleep: what can we do? Curr Opin Anaesthesiol. 2018 Feb;31(1):83-88. doi: 10.1097/ACO.0000000000000538. PMID 29120927
- [Background] Fernandes NM, Nield LE, Popel N, Cantor WJ, Plante S, Goldman L, Prabhakar M, Manlhiot C, McCrindle BW, Miner SE. Symptoms of disturbed sleep predict major adverse cardiac events after percutaneous coronary intervention. Can J Cardiol. 2014 Jan;30(1):118-24. doi: 10.1016/j.cjca.2013.07.009. Epub 2013 Oct 16. PMID 24140074
- [Background] Armstrong KW, Bravo-Iniguez CE, Jacobson FL, Jaklitsch MT. Recent trends in surgical research of cancer treatment in the elderly, with a primary focus on lung cancer: Presentation at the 2015 annual meeting of SIOG. J Geriatr Oncol. 2016 Sep;7(5):368-74. doi: 10.1016/j.jgo.2016.07.004. Epub 2016 Jul 25. PMID 27460994
- [Background] Bolshinsky V, Li MH, Ismail H, Burbury K, Riedel B, Heriot A. Multimodal Prehabilitation Programs as a Bundle of Care in Gastrointestinal Cancer Surgery: A Systematic Review. Dis Colon Rectum. 2018 Jan;61(1):124-138. doi: 10.1097/DCR.0000000000000987. PMID 29219922
- [Background] Minnella EM, Awasthi R, Loiselle SE, Agnihotram RV, Ferri LE, Carli F. Effect of Exercise and Nutrition Prehabilitation on Functional Capacity in Esophagogastric Cancer Surgery: A Randomized Clinical Trial. JAMA Surg. 2018 Dec 1;153(12):1081-1089. doi: 10.1001/jamasurg.2018.1645. PMID 30193337
- [Background] Cho H, Yoshikawa T, Oba MS, Hirabayashi N, Shirai J, Aoyama T, Hayashi T, Yamada T, Oba K, Morita S, Sakamoto J, Tsuburaya A. Matched pair analysis to examine the effects of a planned preoperative exercise program in early gastric cancer patients with metabolic syndrome to reduce operative risk: the Adjuvant Exercise for General Elective Surgery (AEGES) study group. Ann Surg Oncol. 2014 Jun;21(6):2044-50. doi: 10.1245/s10434-013-3394-7. Epub 2014 Mar 27. PMID 24671637
- [Background] Soares SM, Nucci LB, da Silva MM, Campacci TC. Pulmonary function and physical performance outcomes with preoperative physical therapy in upper abdominal surgery: a randomized controlled trial. Clin Rehabil. 2013 Jul;27(7):616-27. doi: 10.1177/0269215512471063. Epub 2013 Feb 12. PMID 23405020
- [Background] Barakat HM, Shahin Y, Khan JA, McCollum PT, Chetter IC. Preoperative Supervised Exercise Improves Outcomes After Elective Abdominal Aortic Aneurysm Repair: A Randomized Controlled Trial. Ann Surg. 2016 Jul;264(1):47-53. doi: 10.1097/SLA.0000000000001609. PMID 26756766
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] Luther A, Gabriel J, Watson RP, Francis NK. The Impact of Total Body Prehabilitation on Post-Operative Outcomes After Major Abdominal Surgery: A Systematic Review. World J Surg. 2018 Sep;42(9):2781-2791. doi: 10.1007/s00268-018-4569-y. PMID 29546448
- [Background] Thomas G, Tahir MR, Bongers BC, Kallen VL, Slooter GD, van Meeteren NL. Prehabilitation before major intra-abdominal cancer surgery: A systematic review of randomised controlled trials. Eur J Anaesthesiol. 2019 Dec;36(12):933-945. doi: 10.1097/EJA.0000000000001030. PMID 31188152
- [Background] Kristjansson SR, Nesbakken A, Jordhoy MS, Skovlund E, Audisio RA, Johannessen HO, Bakka A, Wyller TB. Comprehensive geriatric assessment can predict complications in elderly patients after elective surgery for colorectal cancer: a prospective observational cohort study. Crit Rev Oncol Hematol. 2010 Dec;76(3):208-17. doi: 10.1016/j.critrevonc.2009.11.002. Epub 2009 Dec 14. PMID 20005123
- [Background] Tan KY, Kawamura YJ, Tokomitsu A, Tang T. Assessment for frailty is useful for predicting morbidity in elderly patients undergoing colorectal cancer resection whose comorbidities are already optimized. Am J Surg. 2012 Aug;204(2):139-43. doi: 10.1016/j.amjsurg.2011.08.012. Epub 2011 Dec 16. PMID 22178483
- [Background] Lu J, Cao LL, Zheng CH, Li P, Xie JW, Wang JB, Lin JX, Chen QY, Lin M, Tu RH, Huang CM. The Preoperative Frailty Versus Inflammation-Based Prognostic Score: Which is Better as an Objective Predictor for Gastric Cancer Patients 80 Years and Older? Ann Surg Oncol. 2017 Mar;24(3):754-762. doi: 10.1245/s10434-016-5656-7. Epub 2016 Nov 2. PMID 27807726
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912